CLINICAL TRIAL: NCT04673097
Title: Performance of Different Resin Infiltration Materials on White Spot Lesions: Clinical and Laboratory Assessments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Jumanah Aljishi, Dental intern, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IAU_resin
Record Dates: First submitted 2020-10-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Other: Icon® resin infiltration
- Group 2 (Active Comparator)
  Interventions: Other: MI paste plus
- Group 3 (Active Comparator)
  Interventions: Other: Icon® resin infiltration; Other: MI paste plus

INTERVENTIONS:
Other: Icon® resin infiltration — low viscosity resin that can flow through the pores in the enamel surface
  Arms: Group 1; Group 3
Other: MI paste plus — s a superior form of fluoride ions as it also contains CPP-ACP, enhances mineral release without encouraging the formation of calculus.
  Arms: Group 2; Group 3

SUMMARY:
The study is a clinical controlled trial. Ethical approval will be obtained from Imam Abdulrahman bin Faisal University, Dammam. The study participants will be recruited from the dental hospital and conducted between November 2020 to November 2020. This will be a single-center, randomized, single blinded with a 1:1:1 allocation ratio for the application of Icon® resin infiltration, MI Paste Plus and both treatments

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and able to observe good oral hygiene and attend for the study visits.
* Subjects with ≥1 visible and accessible early caries lesion present.
* No prior white spot lesion treatment utilized except tooth brushing with fluoridated toothpaste.

Exclusion Criteria:

* Active carious lesions
* Facial surface restorations
* Deciduous teeth
* Enamel alteration (fluorosis, opacity, hypocalcification, hypoplasia)
* Intrinsic and extrinsic strains
* Physically and mentally challenged volunteers
* Patients with systemic diseases under medication
* Smokers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2020-12-19 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Color improvements | Change from 0 day, 1 month and 6 months
  Pre-treatment and post-treatment color changing (L*A*B values) of digital photographs using the Commission Internationale de l'Eclairage (CIE) system
Patient self satisfaction | Change from 0 day, 1 month and 6 months
  Post-treatment patient satisfaction using the patient satisfaction scale
Change in lesion status | Change from 0 day, 1 month and 6 months
  Post-treatment change in caries lesion status using ICDAS II
Cracks of enamel. | Change from 0 day, 1 month and 6 months
  Number of cracks assessed by enamel surface analysis via silicone replicas using CLSM
Microbial composition. | Change from 0 day, 1 month and 6 months
  Pre-treatment and post-treatment microbial composition of plaque samples. Samples will be stored at -80 °C until DNA extractions will be performed and run the 16S rRNA sequencing.
Effects on clinical parameter: sensitivity to percussion | Change from 0 day, 1 month and 6 months
  Pre-treatment and post-treatment effects on sensitivity to percussion by end blunted instrument.
esthetic improvement | Change from 0 day, 1 month and 6 months
  Esthetic improvement through objective assessments using a visual analogue
Patient esthetic self perception | Change from 0 day, 1 month and 6 months
  Pre-treatment esthetic self perception by the subjects using questionnaire
change in lesion size | Change from 0 day, 1 month and 6 months
  Pre-treatment and post-treatment white spot lesion size
fracture of enamel. | Change from 0 day, 1 month and 6 months
  Number of fracture assessed by enamel surface analysis via silicone replicas using CLSM
Effects on clinical parameter: prolonged response to hot or cold. | Change from 0 day, 1 month and 6 months
  Pre-treatment and post-treatment effects on response to hot or cold by cold test

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided